CLINICAL TRIAL: NCT00792961
Title: In Vivo Confocal Endomicroscopy During da Vinci Robot Assisted Prostatectomy: Feasibility Study
Brief Title: Real Time Microscopic Imaging During Robot Assisted Prostate Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Delaney (Industry)
Collaborators: Hospital at Westlake (Unknown)
Responsible Party: Sponsor-Investigator, Peter Delaney, Director of Technology, Optiscan Pty Ltd
Organization: Optiscan Pty Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13082008
Record Dates: First submitted 2008-11-16; First posted 2008-11-18 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Robotic surgery; Endomicroscopy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endomicroscopy (Experimental): Endomicroscopy is performed in addition to the patient's indicated robot-assisted prostate surgery
  Interventions: Device: Endomicroscopy

INTERVENTIONS:
Device: Endomicroscopy — Rigid drop-in endomicroscope imaging probe

SUMMARY:
The study involves use of a device called an endomicroscope to obtain high resolution images of microscopic structures during robot-assisted prostate cancer surgery. This feasibility study is largely descriptive, and will use endomicroscopy to document the cellular and architectural appearance of tissue during minimally invasive prostate surgery for later comparison with features seen upon conventional histopathological examination of biopsies or resection specimens.

DETAILED DESCRIPTION:
Prostate surgery requires meticulous dissection around nerves and associated structures such as the bladder, seminal vesicles and vas deferens. Nerve damage during prostatectomy can result in undesirable outcomes such as impotence and urinary incontinence. Robot assisted minimally invasive prostatectomy offers enhanced visualisation of the surgical field. Superior clinical outcomes in terms of length of hospital stay, blood loss, and oncologic margins compared with open surgery are reported. Confocal endomicroscopy provides high resolution subsurface cellular imaging in real time and is already in clinical use in gastroenterology and under investigation in other surgical applications. A potential role exists for confocal endomicroscopy to enhance microscopic nerve identification intra-operatively and guide surgical decision making during robot-assisted prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Males diagnosed with prostate cancer and undergoing da Vinci radical prostatectomy

Exclusion Criteria:

* Patients under 18 years of age
* Patients with allergy or prior adverse reaction to Fluorescein Sodium
* Patients unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Endomicroscopy images captured from prostate and surrounding tissues | During surgery

SECONDARY OUTCOMES:
Comparison with conventional histology from corresponding biopsies or resection specimens | Post-surgery, after pathologist's review

CONTACTS AND LOCATIONS:
Overall Officials: Randy Fagin, MD, Principal Investigator — The Hospital at Westlake Medical Center; Peter Delaney, BSc, Study Director — Optiscan Pty Ltd
Locations (1):
- The Hospital at Westlake Medical Center, Austin, Texas, United States